CLINICAL TRIAL: NCT02490930
Title: A Safety Study of Fingolimod With Radiation and Temozolomide in Newly Diagnosed High Grade Glioma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: J14168; IRB00055036 (Other: JHMIRB)
Record Dates: First submitted 2015-07-02; First posted 2015-07-07 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Glioblastoma; Anaplastic Astrocytoma
Keywords: lymphopenia
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Lymphopenia | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental (Experimental): Five evaluable patients with newly diagnosed high grade gliomas who will undergo standard concomitant radiation and temozolomide followed by adjuvant temozolomide will be accrued to this open-label, single arm, safety study. Oral fingolimod will be given 1 week prior to the initiation of concurrent radiation and temozolomide and will be discontinued immediately upon completion of the six weeks of therapy. Fingolimod will be administered at 0.5 mg every day for the first two weeks. Beginning the third week, they will take fingolimod on Monday, Wednesday and Friday until the end of radiotherapy or until the 28th dose, whichever comes first.
  Interventions: Drug: Fingolimod

INTERVENTIONS:
Drug: Fingolimod — Oral fingolimod will be given 1 week prior to the initiation of concurrent radiation and temozolomide and will be discontinued immediately upon completion of the six weeks of therapy.
  Other Names: Gilenya

SUMMARY:
A recent prospective multicenter study by Dr. Grossman demonstrated that 40% of patients with high grade glioma undergoing radiation and chemotherapy developed severe and persistent lymphopenia (CD4 counts <200 cells/mm3). This lymphopenia lasted for twelve months following radiation treatment and on multivariate analysis was associated with shorter survival. Our group has data that strongly suggests that this lymphopenia is secondary to the inadvertent radiation of circulating lymphocytes as they pass through the radiation beam. Investigators propose the use of FDA approved for multiple sclerosis, fingolimod to signal lymphocytes to leave the circulation prior to the initiation of radiation. It is a functional antagonist of the sphingosine-1-phosphate receptor (S1PR) pathway and prevents lymphocyte egress from secondary lymphoid organs.

Oral fingolimod will be given 1 week prior to the initiation of concurrent radiation and temozolomide and will be discontinued immediately upon completion of the six weeks of therapy. The primary objective is to evaluate if fingolimod can be safely combined with radiation and temozolomide. Secondary endpoint is total lymphocyte counts (TLC) for the proposed study participants. Investigators expect that patients receiving radiation and temozolomide plus fingolimod have a recovery of lymphocyte counts to 80% of baseline within four months, reference to historical control in which sustained lymphopenia lasted for twelve months.

DETAILED DESCRIPTION:
Five evaluable patients with newly diagnosed high grade gliomas who will undergo standard concomitant radiation and temozolomide followed by adjuvant temozolomide will be accrued to this open-label, single arm, safety study. Oral fingolimod will be given 1 week prior to the initiation of concurrent radiation and temozolomide and will be discontinued immediately upon completion of the six weeks of therapy.

The primary objective is to evaluate if fingolimod can be safely combined with radiation and temozolomide. This standard chemoradiation causes 40% of patients to develop severe lymphopenia two months after initiation of therapy. Investigators expect that when this is combined with fingolimod, virtually all patients will have severe lymphopenia two months after beginning treatment. Investigators will determine if these patients who routinely receive pneumocystis jiroveci prophylaxis develop other severe opportunistic infections that would prohibit further evaluation of this novel treatment approach. Primary endpoint is incidence of greater than or equal to Grade III infections attributable to fingolimod-induced lymphopenia defined by the NIH/NCI Common Terminology Criteria for Adverse Events (CTCAE) within four months of starting fingolimod.

The secondary objective is to obtain preliminary information regarding the ability of fingolimod to reduce radiation-related lymphopenia three months after stopping fingolimod. The NIH funded Adult Brain Tumor Consortium (ABTC) followed total lymphocyte and CD4 counts in 96 patients after treatment with radiation and temozolomide. The severe lymphopenia (CD4 count less than 200/mm3) lasted for twelve months in this historical control. Secondary endpoint is total lymphocyte counts (TLC) for the proposed study participants. These will be compared with patient level data on TLC from an historical cohort obtained from the ABTC. Investigators expect that patients receiving radiation and temozolomide plus fingolimod have a recovery of lymphocyte counts to 80% of baseline within four months, reference to historical control in which sustained lymphopenia lasted for twelve months.

Investigators will also obtain laboratory analysis on lymphocyte subtypes and cytokine levels (CD3, CD4, CD8, IL-7, TGF-Beta, etc.). Routine care for high grade gliomas includes weekly Heme-8 and absolute lymphocyte count. Research blood will be obtained at 2 weeks prior to chemoradiation and again at weeks 6, 10, 18, 26 and 46. Patients will be on study for approximately one year.

ELIGIBILITY:
Inclusion Criteria:

* Gender: Male and Female
* Age: Patients must be at least 18 years of age.
* Race: Minorities will be recruited. No exclusion to this study will be based on race.
* Patients must have histologically confirmed high grade astrocytoma, WHO grade III or IV, by pathology.
* Patients' proposed post-operative treatment plan must include standard focal brain irradiation and temozolomide.
* Patients must have a Karnofsky Performance Status > 60 % (i.e. the patient must be able to care for himself/herself with occasional help from others).
* Patients must have normal bone marrow function, with a baseline total lymphocyte count > 1000.
* Patients must be able to provide informed consent.
* Glucocorticoid use is allowed.
* Women of childbearing potential should use effective contraception during and for two months after stopping fingolimod.

Exclusion Criteria:

* Patients must not have received prior radiation therapy, chemotherapy, immunotherapy, therapy with biologic agents or hormonal therapy for their brain tumor.
* Patients must not have recent (within six months) occurrence of myocardial infarction, unstable angina, stroke, transient ischemic attack, decompensated heart failure requiring hospitalization, or Class III/IV heart failure.
* Patients must not have history of or presence of Mobitz Type II 2nd degree or 3rd degree atrioventricular block or sick sinus syndrome, unless patient has a pacemaker.
* Patients must not have baseline QTc interval > 500 ms.
* Patients must not be on treatment with Class Ia or Class III antiarrhythmic drugs.
* Patients must not have a history of macular edema, uveitis or diabetes mellitus.
* Patients must not have elevated liver transaminase levels. Adequate liver function is defined as total bilirubin < 1.5 times upper limit of normal, SGPT (ALT) < 5 times upper limit of normal and serum albumin > 2 g/dL.
* Patients must not have an active infection.
* Patients with known HIV will be excluded.
* Patients with collagen vascular disease are excluded.
* Patients taking immunosuppressive medications (other than dexamethasone) will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Incidence of severe infection attributable to fingolimod-induced lymphopenia | 4 months
  Incidence of greater than or equal to Grade III infections attributable to fingolimod-induced lymphopenia defined by the NIH/NCI Common Terminology Criteria for Adverse Events (CTCAE)

SECONDARY OUTCOMES:
Total lymphocyte counts (TLC) | 4 months
  Total lymphocyte counts (TLC) for study participants compared to TLC for historical control

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Grossman, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No